CLINICAL TRIAL: NCT05514171
Title: PROSPECTIVE REGISTRY OF PATIENTS WITH BORDERLINE AND RESECTABLE PANCREATIC ADENOCARCINOMA IN CATALONIA (PaNLoCat)
Brief Title: Prospective Registry of Patients With Pancreas Adenocarcinoma Resectable and Borderline
Acronym: PaNLoCat
Status: Completed | Type: Observational
Sponsor: Hospital del Mar (Other)
Responsible Party: Principal Investigator, Patricia Sanchez Velazquez, Principal Investigator, Hospital del Mar
Other Study IDs: PaNLoCat_v4
Record Dates: First submitted 2022-08-03; First posted 2022-08-24 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: Chemotherapy Effect; Pancreas Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Neoadyuvant therapy: Patients with borderline or resectable ADK subjected to neoadyuvant therapy
  Interventions: Procedure: Neoadyuvant therapy
- Upfront surgery: Patients with borderline or resectable ADK who undergo upfront surgery

INTERVENTIONS:
Procedure: Neoadyuvant therapy — Patients of group neoadyuvant therapy will receive any chemotherapy treatment before surgery
  Groups: Neoadyuvant therapy

SUMMARY:
Unlike other types of gastrointestinal tumors, there is controversial evidence of the efficacy of neoadjuvant therapy in patients with borderline and resectable adenocarcinoma (ADK) of the pancreas, the objective of this study is to perform a "snapshot" of the usual practice in our setting in terms of neoadjuvant therapy in ADK, both in terms of the different regimens used as well as the results in terms of morbidity, mortality and survival.

Likewise, in a second phase, a prospective registry of patients included in the neoadjuvant regimen for both resectable and borderline ADK diagnosed in Catalonia will be launched, which will provide us with valuable information to try to answer open questions in the context of borderline and resectable ADK treatment.

ELIGIBILITY:
Inclusion Criteria:

* resectable or borderline pancreas ADK
* with or without radiotherapy
* any type of approach
* any type of surgery

Exclusion Criteria:

* locally advanced ADK
* No consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patient who has been diagnosed of ADK resectable or borderline and assessed in a multidiscliplinary tumor board between 2017 and 2021
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Disease free survival | Three years follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital del Mar, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided